CLINICAL TRIAL: NCT05098496
Title: Normative Values of Functional Fitness in Elderly Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: RiphahIU Ayesha Akbar
Record Dates: First submitted 2021-08-20; First posted 2021-10-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Elderly Care; Functional Fitness
Keywords: Normative values; Senior Fitness Test; Functional fitness

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is a multidimensional concept that influences several domains , such as body mass decline, gait ,mobility, balance ,muscle strength ,motor processing ,cognition, nutrition endurance, and physical activity, and its directly related to adverse consequences such as falls ,disability the need for long term care , hospitalization and even mortality. As the elderly have twice as many disabilities and four times as many physical limitations as people less than 60 years of age. There is a need to focus on this demographic shift and Aging population Pakistan increasing double in 2050 hence is has become a new challenge. So, Effective approaches is needed to help older people maintain a healthy and active life. The main objective is to determine reference values of senior fitness test SFT for elderly population. The Senior Fitness Test is a battery of tests for the assessment of the functional fitness of older persons. This test will assess the physiological capacity for carrying out normal daily activities independently and safely without the appearance of fatigue. For this study cross sectional survey will conduct and will use non probability convenience sampling technique , sample size will be 500 both male and female and conducted from Heaven old age homes and Dar ul Khilafa old age home, Lahore. Inclusion criteria includes subject 60 and above , living Subjects 60 years and above, living independently (not community dwelling, hospitals, nurse homes etc ), perform ADLS. Exclusion criteria includes if not willing to participate, any medical contraindication, unable to speech ,functional disability .All the analysis will be carried out on SPSS v -25.

DETAILED DESCRIPTION:
According to the world health organization WHO, the proportion of older people above 60 is growing more rapidly than any other age group. Within this group not everyone reach old age successfully. Although the common rule is that increasing age is related to decreasing well-being and increasing levels of frailty. It is also true that individual with same chronological age can vary in health and functional status . Functional fitness is a way to help people perform daily tasks with ease. It includes exercises that mimic the movements of daily activities. Walking, squatting, bending, pushing, and pulling are examples. Three key elements of functional fitness for seniors are balance, mobility, and strength. Improving these three aspects of physical fitness helps seniors: Maintain a healthy body weight, Reduce the risk of falling, Make activities of daily living easier, Boost emotional health. The discovery of effective interventions to prevent or delay disability in older persons is a public health priority. The geriatric assessment designed to manage frail older people requiring medical care, is responsible for early diagnosis , assessment, treatment, and planning while addressing a person's medical, psychological, social, and functional capabilities.

The purpose of study to highlights age-related differences in physical abilities and the risk for the loss of independence in later life. High walkability of the living environment provides opportunities for physical activity in old age, but among those with physical limitations especially, awareness of environmental facilitators may be needed to promote physical activity. The main objective of this research will be to provide normative values of functional fitness in 60 and above seniors citizens of Pakistan .Research results will enable preparing an effective intervention strategy for maintaining mobility and functional independence of elderly people.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 60 years and above,living independently (not community dwelling, hospitals, nurse homes etc ), moving and performing daily activities independently
2. No medical contraindications to participate in physical fitness tests, with no problems in terms of verbal communication, no physical and cognitive restrictions

Exclusion Criteria:

1. If Participants have any medical contraindications for physical activity programs and to hold medical insurance.
2. Cormobidites ,disability, any cardiac or pulmonary dysfunction (COPD, exercise related exertion etc).
3. Physical condition hindering anthropometric examination (such as immobile patients, contraindication to lifting or amputation of both lower extremities).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Informed consent will be obtained from participants to meet inclusion criteria before including in study.It is a cross sectional study, researcher will find out the normative values of senior citizen by using senior fitness test SFT in both male and female gender 60 or above age .Senior fitness test contains 6 six and before assessment , screening participants either meet inclusion criteria or not and for basic and advanced everyday activities . Anthropometric measurements by BMI body mass index will used. So overall this procedure will contain 45 to 50 minute per participant. All readings of SFT 6 components will be mentioned in table according to gender and age group 60-64yrs ,65-69yrs,70-74yrs,75-79yrs,80-84yrs
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Senior Fitness Test | Day 1
  Functional fitness will be assessed by using the SFT battery includes; 30-Second Chair Stand Test - lower body strength, Arm Curl Test - upper body strength assessment, Chair Sit and-Reach Test - assessment of the flexibility of the lower body, Back Scratch Test - assessment of the flexibility of the upper body, 8-Foot Up-and-Go Test - agility and dynamic balance assessment, 6 - Minute Walk Test - aerobic endurance rating

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naz L, Ghimire U, Zainab A. Behavioral factors associated with utilization of healthcare services among elderly in Pakistan: evidence from a nationally representative survey. BMC Geriatr. 2021 Jan 12;21(1):42. doi: 10.1186/s12877-021-02005-3. PMID 33435874
- [Background] Sabzwari SR, Iqbal R, Fatmi Z, Azam I. Factors associated with geriatric morbidity and impairment in a megacity of Pakistan. PLoS One. 2019 Jun 27;14(6):e0218872. doi: 10.1371/journal.pone.0218872. eCollection 2019. PMID 31247025
- [Background] Clark PG, Blissmer BJ, Greene GW, Lees FD, Riebe DA, Stamm KE. Maintaining exercise and healthful eating in older adults: the SENIOR project II: study design and methodology. Contemp Clin Trials. 2011 Jan;32(1):129-39. doi: 10.1016/j.cct.2010.10.002. Epub 2010 Oct 16. PMID 20955821
- [Background] Chen B, Shin S. Bibliometric Analysis on Research Trend of Accidental Falls in Older Adults by Using Citespace-Focused on Web of Science Core Collection (2010-2020). Int J Environ Res Public Health. 2021 Feb 9;18(4):1663. doi: 10.3390/ijerph18041663. PMID 33572483
- [Background] Ortega FB, Cadenas-Sanchez C, Lee DC, Ruiz JR, Blair SN, Sui X. Fitness and Fatness as Health Markers through the Lifespan: An Overview of Current Knowledge. Prog Prev Med (N Y). 2018 Apr 2;3(2):e0013. doi: 10.1097/pp9.0000000000000013. eCollection 2018 Apr. PMID 32671316